CLINICAL TRIAL: NCT02547103
Title: Efficacy and Safety of Local Application of Chlorhexidine Gluconate Versus Mupirocin Ointment in the Prevention of Peritoneal Dialysis-Related Infection: A Double-Blind, Stratified Randomized Controlled Trial
Brief Title: Chlorhexidine Gluconate Versus Mupirocin Ointment in the Prevention of Peritoneal Dialysis-Related Infection
Acronym: COSMO-PD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Collaborators: Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Principal Investigator, Chidchanok Ruengorn, Faculty of Pharmacy, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: THOR-PD Group
Record Dates: First submitted 2015-09-07; First posted 2015-09-11 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis
Keywords: Chlorhexidine gluconate; Mupirocin ointment; Normal saline; Peritonitis; Peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chlorhexidine gluconate (Experimental): Chlorhexidine gluconate-soaked cloths, clean topical area around catheter exit site with CHG 2% soaked cloths
  Interventions: Other: Chlorhexidine gluconate-soaked cloths
- Normal saline (usual care) (Active Comparator): Normal saline, clean topical area around catheter exit site
  Interventions: Other: Normal saline
- Mupirocin ointment (Active Comparator): Mupirocin ointment 2%, clean topical area around catheter exit site with Mupirocin ointment
  Interventions: Other: mupirocin ointment

INTERVENTIONS:
Other: Chlorhexidine gluconate-soaked cloths
  Arms: Chlorhexidine gluconate
Other: Normal saline
  Arms: Normal saline (usual care)
Other: mupirocin ointment
  Arms: Mupirocin ointment

SUMMARY:
This pilot study aims to evaluate effectiveness, safety, and cost-utility of chlorhexidine gluconate (CHG)-soaked cloths compares to mupirocin ointment and exit site usual care (normal saline) with aseptic technique in prevention of PD-related infection. It is a multicenter, double-blind, stratified randomized controlled trial. Participants will be randomized to three arms mupirocin, usual care, or CHG-soaked cloths in a ratio of 1:1:1. They will be followed up 24 months or completion of PD. The primary outcome is PD-related infection (PD-related peritonitis of exit-site and tunnel infection). Secondary outcomes are infection-related catheter removal and technique failure, nasal and exit-site Staphylococcus aureus colonization, health-related quality of life, mental health, medication adherence, safety, adverse events related to treatments such as skin irritation, rash, etc. Costs include providers and patients expenses. The utility is assessed using the EuroQol (EQ), five-dimensional (5D), five-level (5L) version. The results of this study are anticipated nephrologists and health care professional involving to PD in decision-making for a plan to prevent PD-related infection. In addition, the results will lead to clinical guideline development a prevention of PD-related infection.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is one of renal replacement therapy used for end-stage renal disease. Since 2011, there has been increasing numbers of patients under "PD First" policy of the Thai government. The most common PD related complication is PD-related infection categorized PD-related peritonitis, and exit site and tunnel infection. Although possible to treat PD-related infection, the incidence of technical failure and death due to peritonitis are still high in Thailand. PD-related infections mainly caused by Staphylococcus aureus. To prevent PD-related infection, cleaning with aseptic solvents using aseptic technique and prevent infection by prescribing prophylactic antibiotics are recommended. The International Society for Peritoneal Dialysis (ISPD) has recommended position statement of the regular use of mupirocin ointment around the catheter exits point and apply in nasal cavity. However, there is rising concern of long term use of mupirocin for mupirocin resistance of S. aureus. CHG is antiseptic use in clinical practice. It can coat at least 12 hours on skin and has anti-bacterial covered in both grams negative and positive. Several meta-analysis studies showed effectiveness of CHG in the prevention of hospitals infection i.e. reduces catheter-related sepsis, postoperative infection, and microbial resistance. According to PD-related infection, CHG has very little evidence of its effectiveness. This pilot study aims to evaluate effectiveness, safety, and cost-utility of CHG-soaked cloths compares to mupirocin ointment and exit site usual care (normal saline and povidone-iodine) with aseptic technique in prevention of PD-related infections. It is a multicenter, double-blind, stratified randomized controlled trial. Participants will be randomized to three arms mupirocin, usual care, or CHG-soaked cloths. They will be followed up 24 months or completetion of PD. The primary outcome is PD-related infection (PD-related peritonitis or exit-site and tunnel infection). Secondary outcomes are infection-related catheter removal and technique failure, nasal and exit-site Staphylococcus aureus colonization, health-related quality of life, mental health, medication adherence, safety, adverse events related to treatments such as skin irritation, rash, etc. For cost-utility analysis, costs include providers and patients expenses. The Utility is assessed using EQ-5D-5L.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end-stage renal disease who were undergoing peritoneal dialysis; either continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dialysis (APD)

Exclusion Criteria:

1. History of psychological illness or condition that interferes with the ability to understand or comply with the requirements of the study
2. Recent (within 1 month) exit-site or tunnel infection, or peritonitis
3. Known hypersensitivity to, or intolerance of, chlorhexidine gluconate, or mupirocin
4. Current or recent (within 1 month) treatment with antibiotics administered by any route
5. Nasal carriage of mupirocin-resistant Staphylococcus aureus or chlorhexidine-resistant S. aureus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of PD-related infections | 24 months
  Peritonitis or exit-site and tunnel infection

SECONDARY OUTCOMES:
Incidence of infection-related catheter removal | 24 months
  Peritonitis or exit-site and tunnel infection-related catheter removal
Incidence of hospitalization due to PD-related infection | 24 months
Incidence of PD technical failure (change of modal of dialysis) | 24 months
  change of modal of dialysis
Incidence of death due to PD-related infection | 24 months
  Death due to peritonitis or exit-site and tunnel infection
Rate of Staphylococcus aureus colonization | 24 months
  Incidence of nasal or exit-site S. aureus colonization
Changes in health-related quality of life | 24 months
  Using the Kidney Disease Quality of Life-36 (KDQOL-36), EuroQoL-5 dimension-5 level (EQ-5D-5L)
Number of participants with depression | 24 months
  Using the Beck Depression Inventory II (BDI-II)
Changes in medication adherence | 24 months
  Using (i) directly observed to record the use of investigational medicinal products via return plastic sachets and ointment tubes; (ii) global rating on medication adherence by visual analog scale; and (iii) Medication-taking behavior measure for Thai patients (MTB-Thai questionnaire
Total healthcare costs | 24 months
  Direct medical costs, direct non-medical costs, and indirect costs
Incidence of skin reactions | 24 months

OTHER OUTCOMES:
Safety profiles | 24 months
  Safety of investigational medicinal products related to potential harm (e.g. participant survival, hospitalization, and emergency visit)

CONTACTS AND LOCATIONS:
Overall Officials: Chidchanok Ruengorn, Study Director — Faculty of Pharmacy CMU
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nochaiwong S, Ruengorn C, Noppakun K, Panyathong S, Dandecha P, Sood MM, Saenjum C, Awiphan R, Sirilun S, Mongkhon P, Chongruksut W, Thavorn K; Thai Renal Outcomes Research (THOR) Investigators. Comparative Effectiveness of Local Application of Chlorhexidine Gluconate, Mupirocin Ointment, and Normal Saline for the Prevention of Peritoneal Dialysis-related Infections (COSMO-PD Trial): a multicenter randomized, double-blind, controlled protocol. Trials. 2019 Dec 19;20(1):754. doi: 10.1186/s13063-019-3953-8. PMID 31856900
- See also: Faculty of Pharmacy, Chiang Mai University — http://www.pharmacy.cmu.ac.th